CLINICAL TRIAL: NCT07084116
Title: Evaluation of Tretinoin Cream on the Integrity of Aged Forearm Skin: an Open-label Within-subject Randomized Study
Brief Title: Evaluation of Tretinoin Cream on the Integrity of Aged Forearm Skin
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kristin M. Nord, Primary Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 77594
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Skin Tear; Solar Purpura; Dermatoporosis
Keywords: skin tear; thin skin
MeSH Terms: interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: Patients will either apply the test cream (tretinoin 0.1% cream) to the right or left arm and a bland cream (placebo) to the other - they will be randomized to right or left arm based on handedness (dominant vs non-dominant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm participants apply tretinoin (LEFT or RIGHT) (Active Comparator): Participants will apply tretinoin 0.1% cream nightly for 6 months.
  Interventions: Drug: Tretinoin 0.1% cream; Drug: Bland cream (non-drug)
- Arm participants apply bland cream (not treatment) (LEFT or RIGHT) (Placebo Comparator): Participants apply bland cream to the other arm nightly as a placebo.
  Interventions: Drug: Bland cream (non-drug)

INTERVENTIONS:
Drug: Tretinoin 0.1% cream — Tretinoin 0.1% cream formulation.
  Other Names: Bland cream (non-medicated)
  Arms: Arm participants apply tretinoin (LEFT or RIGHT)
Drug: Bland cream (non-drug) — Bland cream formulation.

SUMMARY:
The purpose of this research is to determine whether once nightly application of tretinoin 0.1% cream to forearm skin reduces the frequency of skin tears and bruising (solar purpura), and changes skin thickness over a period of 6 months.

DETAILED DESCRIPTION:
Easy bruising and tearing of forearm skin is common with aging and can cause activity restriction, infection, and pain. Chronic exposure to UV light from the sun causes skin thinning and loss of supportive collagen over time. Thin skin tears easily and blood vessels normally protected by collagen rupture, causing bruises. Tretinoin is a prescription vitamin A cream that has been shown to increase skin thickness and collagen. Tretinoin is FDA approved for treatment of acne. We are trying to figure out if putting tretinoin cream on the forearms of adults with thin skin prevents skin tears and bruising.

This research study is looking for 30 people with a history of skin tears in the United States. The VA Palo Alto expects to enroll 30 research study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult (55+)
* History of skin tears, at least 2 in the past month
* History of skin bruising (solar purpura)
* Ambulatory
* Able to apply topical medication to oneself

Exclusion Criteria:

* <55 years old)
* Pregnant or breastfeeding
* History of allergy to tretinoin
* History of atopic dermatitis, psoriasis, bullous skin disease, cutaneous lupus, or cutaneous T cell lymphoma.
* Planned cutaneous surgery on either forearm in the next 6 months
* Use of any topical medication on the forearms within past month
* Current or anticipated phototherapy of the forearms in the next 6 months
* Current or anticipated chemotherapy within the next 6 months
* Use of oral steroids within past month
* Current or prior isotretinoin therapy within past 6 months
* AV fistula of the arm

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of skin tears. | 6 months.
Change in epidermal (top layer of skin) thickness. | 6 months.

SECONDARY OUTCOMES:
Change in percent of skin on the arms involved by solar purpura (bruising). | 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto VA Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
Restriction as part of monitoring agreement.

REFERENCES:
- [Background] Sitohang IBS, Makes WI, Sandora N, Suryanegara J. Topical tretinoin for treating photoaging: A systematic review of randomized controlled trials. Int J Womens Dermatol. 2022 Mar 25;8(1):e003. doi: 10.1097/JW9.0000000000000003. eCollection 2022 Mar. PMID 35620028